CLINICAL TRIAL: NCT00942604
Title: A Multi-center, Randomized, Parallel Group, Double-blind, Vehicle-controlled Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel, 0.05%, In Patients With Actinic Keratoses on Non-head Locations (REGION-Ib)
Brief Title: A Multicenter Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel When Used to Treat Actinic Keratoses (AKs) on the Non Head Locations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEP005-028
Record Dates: First submitted 2009-07-19; First posted 2009-07-21 (Estimated); Results first posted 2012-03-19 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2013-11

CONDITIONS: Actinic Keratoses
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP005 (ingenol mebutate) Gel (Active Comparator): PEP005 (ingenol mebutate) Gel 0.05% once daily for 2 consecutive days
  Interventions: Drug: PEP005 (ingenol mebutate) Gel
- Vehicle gel (Placebo Comparator): Vehicle gel once daily for 2 consecutive days
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: PEP005 (ingenol mebutate) Gel — two day treatment
  Arms: PEP005 (ingenol mebutate) Gel
Drug: Vehicle gel — two day treatment
  Arms: Vehicle gel

SUMMARY:
The purpose of this study is to determine whether topical application of PEP005 is effective for the treatment of actinic keratoses.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age.
* Female patients must be of:
* Non-childbearing potential;
* Childbearing potential, provided negative serum and urine pregnancy test and using effective contraception.
* 4 to 8 AK lesions on non-head locations.

Exclusion Criteria:

* Cosmetic or therapeutic procedures within 2 weeks and within 2 cm of the selected treatment area.
* Treatment with immunomodulators, or interferon/ interferon inducers or systemic medications that suppress the immune system within 4 weeks.
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy within 8 weeks and 2 cm of treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Burke Pharmaceutical Research, Hot Springs, Arizona
  - Skin Surgery Medical Group Inc., San Diego, California
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Skin Specialists, PC, Omaha, Nebraska
  - Karl G. Heine Dermatology, Henderson, Nevada
  - Group Health Associates, Cincinnati, Ohio
  - DermResearch, Inc., Austin, Texas
  - Suzanne Bruce and Associates, PA, The Center for Skin Research, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Dermatology Associates of Tyler, Tyler, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education and Research Foundation, Lynchburg, Virginia
  - Virginia Clinical Research, Inc, Norfolk, Virginia

REFERENCES:
- [Derived] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- See also: Food and Drug Authority — http://www.fda.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period was 22 July 2009 (first patient randomized) to 14 October 2009 (last patient completed Day 57).
Period: Overall Study
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Started | 100 | 103
Completed | 98 | 99
Not Completed | 2 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Patient relocation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel | Total
Number analyzed (Participants) | 100 | 103 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 52 | 100
  >=65 years | 52 | 51 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 35 | 76
  Male | 59 | 68 | 127
Region of Enrollment [Number; unit: participants]
  United States | 100 | 103 | 203

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete Clearance of Actinic Keratoses (AK) Lesions
Description: Proportion of Patients with Complete Clearance of the treatment field defined as no clinically visible Actinic Keratoses (AK) lesions in the selected treatment area
Time Frame: 57 days
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Number analyzed (Participants) | 100 | 103
participants | 42 | 5
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel vs Vehicle Gel; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Proportion of Patients With Partial Clearance of Actinic Keratoses (AK) Lesions
Description: Proportion of patients with Partial Clearance defined as ≥ 75 % reduction in the number of Actinic Keratoses (AK) lesions identified at baseline in the treatment area
Time Frame: 57 days
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Number analyzed (Participants) | 100 | 103
participants | 55 | 7
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel vs Vehicle Gel; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 57 days
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 2/100 | 2/103
Other Adverse Events (participants affected / at risk) | 18/100 | 1/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEP005 (Ingenol Mebutate) Gel (N=100) | Vehicle Gel (N=103)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEP005 (Ingenol Mebutate) Gel (N=100) | Vehicle Gel (N=103)
Application site pruritus (Skin and subcutaneous tissue disorders) | 16 | 0
Application site irritation (Skin and subcutaneous tissue disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For US sites: The institution and investigator agree not to publish the results of this study without prior written consent of the Sponsor. As used herein, the term "publish" shall include oral presentations,written abstracts, written manuscripts, etc.